CLINICAL TRIAL: NCT07077096
Title: Diagnostic Utility of Pleural Infection-specific Multiplex PCR Panel to Identify Causative Microorganisms in Pleural Infection
Brief Title: Diagnostic Utility of Pleural Infection-specific Multiplex PCR Panel
Acronym: PRISM
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: PRISM
Record Dates: First submitted 2025-07-03; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pleural Infection
Keywords: Parapneumonic effusion; Pleural effusion; Empyema
MeSH Terms: conditions — Pleural Effusion; Empyema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pleural fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pleural infection: Patients with pleural infection
  Interventions: Diagnostic Test: PRISM PCR panel; Diagnostic Test: Conventional bacterial culture
- Non-pleural infection: Patients without pleural infection
  Interventions: Diagnostic Test: PRISM PCR panel; Diagnostic Test: Conventional bacterial culture

INTERVENTIONS:
Diagnostic Test: PRISM PCR panel — Comparing the diagnostic accuracy between conventional bacterial culture and multiplex PCR on diagnosing pleural infection
Diagnostic Test: Conventional bacterial culture — Comparing the diagnostic accuracy between conventional bacterial culture and multiplex PCR on diagnosing pleural infection

SUMMARY:
Pleural effusion is a common cause of hospitalization. Pleural infection ranked third among the pleural effusions requiring hospitalization in the United States. Pleural infection, including complicated parapneumonic effusion and empyema, is associated with a 30-day mortality of 10%. Approximately 20-57% of patients with pneumonia have an associated pleural effusion at presentation, of which 5-7% progress to pleural infection. Analyses of several nation-wide healthcare databases in the United States, France and the United Kingdom have showed an increasing incidence of pleural infection in the past decade.

Adequate antibiotic coverage and fluid drainage are the two pillars of treatment for pleural infection. The empirical use of antibiotics should be based on the local spectrum of causative microorganisms and the source of infection. Subsequent targeted antibiotic regimen can be guided by the culture results and sensitivity pattern of the cultured microorganisms. The use of blood culture bottles as the transfer medium can improve the culture positivity from 30-40% to 60%. An explorative study of culturing pleural tissue can increase the microbiological yield from 20% to 45%. Despite these methods, the culture positivity rates are far from 100% although clinical evidence of pleural infection. Peripheral blood cultures may occasionally be the only positive source of culture (12%). Occasionally, complicated malignant pleural effusion (MPE) can mimic pleural infection, by sharing similar biochemical features of high neutrophil counts and lactate dehydrogenase in the pleural fluid. This would subject the patients with MPE to unnecessary prolonged course of antibiotic and delay of chemotherapy. Prolonged course of broad-spectrum antibiotics (BSA) is commonly required for culture-negative pleural infection or MPE with complicated features, but it could lead to various antibiotic-related adverse events, including kidney and liver injuries, opportunistic infections (e.g. Clostridioides difficile colitis). These are clinical unmet needs of identifying causative microorganisms in pleural infection.

The application of multiplex bacterial polymerase chain reaction (PCR) panel has transformed the care of patients with respiratory infection. Incorporating multiplex bacterial PCR test of bronchoalveolar lavage in hospitalized patients with pneumonia at risk of Gram-negative bacterial infection can significantly shorten the duration of inappropriate antibiotic therapy. For patients with suspected lower respiratory tract infection, this platform allows early antibiotic adjustment (faster antibiotic escalations for Gram-negative or Gram-positive bacteria, and faster antibiotic de-escalations directed at Gram-positive bacteria). The use of multiplex PCR panel designed for pneumonia has been applied to patients with parapneumonic effusion with successful identification of non-culturable microorganism. However, the use of pneumonia multiplex PCR panels has not been fully validated in the clinical management of pleural infection. More importantly, these panels only detect common microorganisms included on their panels specifically designed for pneumonia. Therefore, a dedicated pleural infection-specific multiplex (PRISM) PCR panel is required to enhance the identification for microorganisms in patients presenting with pleural infection.

A syndromic real-time PCR panel for diagnosing community-acquired pleural infection has been established by a Norway group, with its components constructed based on the next-generation sequencing results using prior pleural infection samples. Their panel showed a higher diagnostic sensitivity than that of conventional culture-based methods. For bacterial species included in the PCR panel, it had a sensitivity of 99.5%. However, it lacks clinical performance data and may not be applicable in the South-East Asian region as the microbiological spectrum of pleural infection differs geographically, with pneumococci and viridans streptococci the most commonly reported isolates from tropical and temperate regions, respectively. Therefore, a PRISM PCR panel dedicated for South-East Asian population is highly warranted. The investigators has developed a PRISM PCR panel dedicated for local population. The investigators hypothesize that this new PRISM PCR panel has higher diagnostic sensitivity than conventional culture-based methods in identifying causative microorganisms in prospectively collected real-world pleural fluid specimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for new-onset pleural effusion requiring thoracentesis
* Aged 18 years old or above

Exclusion Criteria:

* History of tuberculous pleuritis and bacterial pleural infection in the ipsilateral pleural space
* History of intrapleural therapy (including talc and fibrinolytic) in the ipsilateral pleural space
* History of surgical decortication or pleurodesis in the ipsilateral pleural space
* Eczematous or infected cutaneous conditions at the site of planned pleural procedure that may increase the risk of contamination during the procedure
* Failed to obtain informed consent due to the patient's refusal or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pleural infection will be recruited as positive control. Patients without pleural infection will be recruited as negative control.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic sensitivity and specificity of the PRISM PCR panel | 24 months
  The diagnostic performance (sensitivity and specificity ) of the PRISM PCR panel and conventional bacterial culture in diagnosing pleural infection

SECONDARY OUTCOMES:
the effect of antibiotic on the diagnostic sensitivity and specificity of PRISM PCR panel | 24 months
  Evaluation of the effect of time difference between intiation of antibiotic and pleural fluid aspiration on the diagnostic accuracy (sensitivity and specificity) of PRISM PCR panel in diagnosing pleural infection
the effect of pleural fluid pH on the diagnostic sensitivity and specificity of PRISM PCR panel | 24 months
  Evaluation of the effect of pleural fluid pH on the diagnostic accuracy (sensitivity and specificity) of PRISM PCR panel in diagnosing pleural infection

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No